CLINICAL TRIAL: NCT03511573
Title: ROLIVER - Prospective Cohort for the Identification of Liver Microbiota
Acronym: ROLIVER
Status: Completed | Type: Observational
Sponsor: Tîrgu Mureș Emergency Clinical County Hospital, Romania (Other)
Responsible Party: Principal Investigator, Radu Mircea Neagoe, Associate Professor, Tîrgu Mureș Emergency Clinical County Hospital, Romania
Other Study IDs: TirguMECCH
Record Dates: First submitted 2018-04-18; First posted 2018-04-30 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: To Generate Microbial Hypotheses Putatively Responsible for the Onset of Liver Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bariatric and other laparoscopic surgery — We have obtained liver samples during laparoscopic surgical procedures in the majority of cases. The majority of laparoscopic procedures were sleeve gastrectomies performed for morbid obesity as a primary restrictive procedure; in 5 cases the liver biopsies were performed during laparoscopic cholecystectomies.

SUMMARY:
The existence of an adipose tissue microbiota causally involved in the triggering of a low grade inflammation could resemble what observed in liver fibrosis. To generate microbial hypotheses putatively responsible for the onset of liver fibrosis we sequenced the 16SrDNA gene from liver biopsies from 36 obese patients (ROLIVER cohort) and describe an original mathematical approach to decipher signatures of early stage of liver fibrosis F0, F1, F2.

DETAILED DESCRIPTION:
Liver diseases and notably fibrosis are featured by a gut microbiota dysbiosis with a large diversity. Classical statistical analyses does not allow to discriminate between the different low score of liver fibrosis F0,F1,F2. The existence of an adipose tissue microbiota causally involved in the triggering of a low grade inflammation could resemble what observed in liver fibrosis. To generate microbial hypotheses putatively responsible for the onset of liver fibrosis we sequenced the 16SrDNA gene from liver biopsies from 36 obese patients (ROLIVER cohort) and describe an original mathematical approach to decipher signatures of early stage of liver fibrosis F0, F1, F2. We identified that Protebacteria as the main phyla in liver with Pseudomonadaceae and Proteobacteriaceae families representing ~60% of the 16SrDNA gene diversity. While primary component analyses were unable to discriminate between the three groups the partial least square discriminant analysis appears as a powerful tool to identify signatures predictive for each group. We further constructed a matrix of interacting OTU clusters surrounding early scores of liver fibrosis. Eventually, we applied the tfidf approach to exemplify the rare variables which could be carrying some information suitable to refine the diagnosis. Altogether, we here propose a mathematical approach suitable for precise identification of bacteria putatively involve in the progressive development of liver fibrosis that represent hence a new therapeutic opportunity.

ELIGIBILITY:
Inclusion Criteria:

* bariatric patients
* morbid obesity patients

Exclusion Criteria:

* serious chronic associated illness (heart failure, cirrhosis, panhypopituitarism or autoimmune diseases), consumption of alcohol (> 20 g ethanol intake per day), related use of medication (use of laxatives, fiber supplements or probiotics in the previous 6 weeks), inflammatory disorders and use of immunomodulatory drugs. Other exclusion criteria were: history of bariatric surgery, use of anti-obesity drugs in the previous 3 months, recent (last 2 months) or on-going antibiotic use, excessive use of vitamin D supplementation; active or recent (last 3 months), participation in a weight loss program or weight change of 3 kg during the past 3 months, pregnant or planning pregnancy within 6 months or breastfeeding women, drug abuse, and other reasons identified by the Investigator.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Eligible participants were males or females with a BMI over 35 and comorbidities or over 40.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
a positive or a negative linear regression between 16SrDNA sequences and liver fibrosis scores | 36 months
  the frequency of some 16SrDNA in the liver should be positively or negatively correlated with the score of liver fibrosis

IPD SHARING:
Plan to Share IPD: Undecided